CLINICAL TRIAL: NCT02106624
Title: The Efficacy and Safety of High Nitrogen Intake in Critically Ill Patients: a Randomized and Controlled Trial
Brief Title: A Trial to Assess the Effect of High Nitrogen Intake in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Ming Zhong, Associate Professor of Division of Critical Care Medicine, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HiNiCi
Record Dates: First submitted 2014-03-30; First posted 2014-04-08 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Critically Ill
Keywords: mechanical ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Nitrogen (Experimental): In this arm, daily nitrogen supply is as much as 2.5-3.0 g per kilogram (lean mass weight)
  Interventions: Other: nitrogen supply
- conventional nitrogen (Active Comparator): In this arm, daily nitrogen supply is 1.2-1.5g per kilogram (lean mass weight) as recommended by ESPEN guideline
  Interventions: Other: nitrogen supply

INTERVENTIONS:
Other: nitrogen supply — Nitrogen supply could be administered through amino acid in parenteral nutrition, proteins in enteral nutrition.

SUMMARY:
The patients with sepsis are in high risk of malnutrition, which could contribute to infection, difficulty in weaning from ventilators. The investigators speculate whether nutrition therapy with high nitrogen could attenuate the malnutrition status and improve the outcome in these sepsis patients. In this prospective Randomized Controlled Trial, the investigators aim to compare high nitrogen intake with conventional nitrogen supply which were recommended in guidelines.

ELIGIBILITY:
Inclusion Criteria:

* need mechanical ventilation for more than 2 days
* mean blood pressure more than 60mmHg
* predicted ICU stay more than 7 days
* tolerance of parenteral or enteral nutrition

Exclusion Criteria:

* irreversible status of primary disease
* any history of malnutrition before enrollment
* history of steroid cortisol administration
* severe liver dysfunction (Child-Pugh Score C)
* pregnancy
* refuse to enrollment
* re-admission to ICU and has been enrolled during former admission to ICU

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 28 days
all cause mortality | 90 days

SECONDARY OUTCOMES:
duration on ventilators | patients enrolled will be followed for the duration of mechanical ventilation, an expcected average of 4 weeks
ICU stay | patients enrolled will be followed for length of ICU stay, an expected average of 6 weeks
infection incidence rate | 28 days
  Details of infection includes pneumonia, catheter-related blood stream infection, urinary tract infect, et al. Diagnosis of infection accords to symptoms, lab tests, imaging measurements and bacterial cultures.
Liver function and renal function | on 1st. day, 3rd. day, 7th. day, 14th. day, 21st. day, 28th. day after enrollment
  Liver function is assessed through serum bilirubin and liver enzyme, renal function is assessed through serum urea nitrogen and creatinine.
diameter of midpoint of musculus rectus femoris | on 28th. day or endpoint of the trial
  diameter of the muscle is measured with percutaneous ultrasound
serum concentration of albumin, pre albumin, retinaldehyde binding protein, transferrin | on 7th. day , 14th. day, 21st. day, 28th. day after enrollment
change of body composition | on 7th.day, 14th.day, 21st.dat, 28th.day after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Critical Care Medicine: Zhongshan Hospital, Shanghai, Shanghai Municipality, China